CLINICAL TRIAL: NCT02164292
Title: Associating Liver Partition and Portal Vein Ligation for Staged Hepatectomy (ALPPS): Safety, Feasibility and Efficacy at a Single Center
Brief Title: ALPPS: Safety, Feasibility and Efficacy at a Single Center
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 1942
Record Dates: First submitted 2014-06-11; First posted 2014-06-16 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Locally Advanced Malignant Liver Disease
Keywords: Liver tumor; ALPPS; Two-stage hepatectomy; Morbidity; Hypertrophy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hypertrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALPPS group: Patients with small future liver remnant who are operated with the "Associating Liver Partition and Portal vein ligation for Staged hepatectomy" approach
  Interventions: Procedure: ALPPS

INTERVENTIONS:
Procedure: ALPPS — Associating Liver Partition and Portal vein ligation for Staged hepatectomy

SUMMARY:
The possibility to achieve a curative resection in patients with liver malignancies is limited by the future liver remnant (FLR). The Associating Liver Partition and Portal vein ligation for Staged hepatectomy (ALPPS) approach has recently been introduced as a revolutionary strategy to achieve resectability by inducing a rapid and large FLR hypertrophy. However, the possibility of achieving a short-term hypertrophy and high resectability rates has been counteracted in most published series by an increased risk of morbidity and mortality.The aim of this study was to evaluate the results with the ALPPS procedure in a single high-volume HPB center, with special emphasis in the safety and feasibility of this new 2-stage strategy. The aim of the present study was to assess the safety, feasibility and efficacy of ALPPS in a single high-volume hepatobiliary center.

DETAILED DESCRIPTION:
Complete resection of liver malignancies remains as the best treatment to offer the possibility of long-term survival or cure. At diagnosis, many patients have locally advanced disease that often precludes a curative resection. During the past two decades, a better assessment of resectability through modern imaging techniques along with new multimodal therapies and the introduction of modern chemotherapy regimens have allowed to increase the pool of candidates for surgical treatment in patients with locally advanced disease. The current principles for safe liver resections focus mainly on the liver parenchyma that remains after resection rather than the liver resected. In fact, one of the main conditioning factors of posthepatectomy liver failure (PHLF) is the amount and quality of future liver remnant (FLR). The induction of hypertrophy of healthy parenchyma using either portal vein embolization (PVE) or ligation (PVL), in the setting of 1-stage or 2-stage liver resections, is nowadays considered the standard of care for patients with locally advanced liver tumors and small FLR.2,5-8 However, the need for long intervals between interventions (6-12 weeks), results in resectability rates that rarely exceed 60-80%.

In 2012, Schnitbauer et al introduced a novel 2-stage technique that allowed tumor resection in 25 patients from 5 German centers with marginally resectable or primarily nonresectable disease by means of a rapid and large FLR hypertrophy. This technique was later popularized with the acronym ALPPS for "Associating Liver Partition and Portal Vein Ligation for Staged Hepatectomy". The promising preliminary results obtained with this new surgical proposal in terms of hypertrophy and the possibility of challenging the previous methods generated a pronounced reaction in the surgical community world-wide that has rarely been seen in the history of hepato-pancreato-biliary (HPB) surgery. However, the possibility of achieving a short-term hypertrophy and high resectability rates has been counteracted in most published series by an increased risk of morbidity and mortality. The aim of this study was to evaluate the results with the ALPPS procedure in a single high-volume HPB center, with special emphasis in the safety and feasibility of this new 2-stage strategy.

Data for all patients undergoing 2-stage hepatectomies with the ALPPS approach at the HPB Surgery Section of the Hospital Italiano de Buenos Aires between June 2011 and April 2014 was analyzed on an intention to treat basis. Patient demographics, clinical characteristics (body mass index, anesthesiological risk score, Charlson comorbidity index, preoperative chemotherapy), tumor type, surgical details, FLR hypertrophy, postoperative liver function, postoperative complications, length of hospital stay and survival were analyzed.

Regarding the surgical procedure, during the first stage a complete tumor resection (clean-up) of the FLR is performed if bilateral disease was present, either trough anatomical or atypical resections. Subsequently, the portal vein of the diseased hemi-liver (DH) is divided and either total (up to the inferior vena cava) or partial (up to the middle hepatic vein) parenchymal transection using the Cavitron Ultrasonic Surgical Aspirator (CUSA; Valley Lab, Boulder, CO, USA) is carried out. At the end of the first stage, the DH is either wrapped in a plastic bag or a plastic sheath placed between the cut surfaces. Once volumetric CT analysis demonstrated enough FLR hypertrophy and provided the patient is in good condition, the second stage is carried out the next available operative day resecting the DH. The type of liver resections performed were defined using the Brisbane 2000 nomenclature.

ELIGIBILITY:
Inclusion Criteria:

* Patients with marginally resectable or primarily non-resectable locally advanced liver tumors
* Insufficient FLR either in volume or quality

Exclusion Criteria:

* Unresectable liver metastases in the future liver remnant or unresectable extrahepatic metastases
* Severe portal hypertension
* High anesthesiological risk
* Unresectable primary tumor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-Volume University Hospital population
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety of the procedure defined as the incidence of postoperative complications and mortality | within the first 90 days after the first stage
  Ocurrence of any postoperative complication or mortality considering the Dindo-Clavien classification of surgical complications
Feasibility of the procedure defined as percentage of patients that complete both surgical stages. | within 4 months after the first stage
  Percentage of patients that finally arrive to the 2nd stage of the ALPPS approach

SECONDARY OUTCOMES:
Efficacy of the procedure defiend as the percentage of patients who achieve a sufficient future liver remnant hypertrophy | within 10 days after the first stage
  Achievement of sufficient short-term hypertrophy of the future liver remnant (FLR). Sufficiency was defined as a FLR >0.5% of body weight or >25% of standardized total liver volume in case of healthy liver parenchyma, or >0.8% and 40% in case of diseased parenchyma.
Disease-free survival and overall survival | 1 and 2 years
  Disease free survival was the time that a patient remained alive and without evidence of disease from the second stage. Overall survival was the time from the first stage to patient death.
Risk factors for morbidity | within 3 month after the first stage
  To identify clinical or operative risk factors of postoperative complications
Risk factors for a reduced kinetic growth rate of the future liver remnant (<35 cc/day) | within 3 months after the first stage
  To identify clinical or operative risk factors or a reduced kinetic growth rate of the future liver remnant (<35 cc/day)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo de Santibañes, MD, PhD, Study Director — General Surgery Service, Hospital Italiano de Buenos Aires. Argentina
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Background] Agrawal S, Belghiti J. Oncologic resection for malignant tumors of the liver. Ann Surg. 2011 Apr;253(4):656-65. doi: 10.1097/SLA.0b013e3181fc08ca. PMID 21475004
- [Background] Clavien PA, Petrowsky H, DeOliveira ML, Graf R. Strategies for safer liver surgery and partial liver transplantation. N Engl J Med. 2007 Apr 12;356(15):1545-59. doi: 10.1056/NEJMra065156. No abstract available. PMID 17429086
- [Background] Mise Y, Sakamoto Y, Ishizawa T, Kaneko J, Aoki T, Hasegawa K, Sugawara Y, Kokudo N. A worldwide survey of the current daily practice in liver surgery. Liver Cancer. 2013 Jan;2(1):55-66. doi: 10.1159/000346225. PMID 24159597
- [Background] Schnitzbauer AA, Lang SA, Goessmann H, Nadalin S, Baumgart J, Farkas SA, Fichtner-Feigl S, Lorf T, Goralcyk A, Horbelt R, Kroemer A, Loss M, Rummele P, Scherer MN, Padberg W, Konigsrainer A, Lang H, Obed A, Schlitt HJ. Right portal vein ligation combined with in situ splitting induces rapid left lateral liver lobe hypertrophy enabling 2-staged extended right hepatic resection in small-for-size settings. Ann Surg. 2012 Mar;255(3):405-14. doi: 10.1097/SLA.0b013e31824856f5. PMID 22330038
- [Background] de Santibanes E, Clavien PA. Playing Play-Doh to prevent postoperative liver failure: the "ALPPS" approach. Ann Surg. 2012 Mar;255(3):415-7. doi: 10.1097/SLA.0b013e318248577d. No abstract available. PMID 22330039
- [Background] Shindoh J, Vauthey JN, Zimmitti G, Curley SA, Huang SY, Mahvash A, Gupta S, Wallace MJ, Aloia TA. Analysis of the efficacy of portal vein embolization for patients with extensive liver malignancy and very low future liver remnant volume, including a comparison with the associating liver partition with portal vein ligation for staged hepatectomy approach. J Am Coll Surg. 2013 Jul;217(1):126-33; discussion 133-4. doi: 10.1016/j.jamcollsurg.2013.03.004. Epub 2013 Apr 28. PMID 23632095
- [Background] Schadde E, Ardiles V, Slankamenac K, Tschuor C, Sergeant G, Amacker N, Baumgart J, Croome K, Hernandez-Alejandro R, Lang H, de Santibanes E, Clavien PA. ALPPS offers a better chance of complete resection in patients with primarily unresectable liver tumors compared with conventional-staged hepatectomies: results of a multicenter analysis. World J Surg. 2014 Jun;38(6):1510-9. doi: 10.1007/s00268-014-2513-3. PMID 24748319
- [Background] Torres OJ, Fernandes Ede S, Oliveira CV, Lima CX, Waechter FL, Moraes-Junior JM, Linhares MM, Pinto RD, Herman P, Machado MA. Associating liver partition and portal vein ligation for staged hepatectomy (ALPPS): the Brazilian experience. Arq Bras Cir Dig. 2013 Jan-Mar;26(1):40-3. doi: 10.1590/s0102-67202013000100009. English, Portuguese. PMID 23702869
- See also: Worldwide registry of Associating Liver Partition and Portal vein Ligation for Staged hepatectomy (ALPPS) — http://www.alpps.net